CLINICAL TRIAL: NCT05308706
Title: Double-blind Randomized Placebo-controlled Trial of the Efficacy of the Apollo System for Children With ADHD
Brief Title: Efficacy of the Apollo System for Children With ADHD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Michigan State University (Other)
Collaborators: The Board of Medicine (Other)
Responsible Party: Principal Investigator, Matthew B. Pontifex, Ph.D., Associate Professor, Michigan State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: STUDY00005951
Record Dates: First submitted 2022-03-24; First posted 2022-04-04 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: ADHD; Inhibition; Vibrational therapy
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Inhibition, Psychological

STUDY DESIGN:
Intervention Model Description: All participants receive an Apollo System device. However, participants are randomly assigned to receive a device that uses the current pattern of vibrations as in the commercial Apollo System device or receive a device that uses an ultra-low frequency pattern of vibrations (sham device).
Who Masked: Participant, Investigator
Masking Description: Double blind, sham/placebo controlled trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Commercial Apollo System Device (Experimental): The active experimental group received the commercial Apollo System device.
  Interventions: Device: 8 weeks of home based use.
- Sham Apollo System Device (Sham Comparator): The control experimental group received a sham/placebo device that is identical to the commercial Apollo System device but uses an ultra-low (i.e., effectively zero) frequency pattern of vibrations.
  Interventions: Device: 8 weeks of home based use.

INTERVENTIONS:
Device: 8 weeks of home based use. — Use of the devices for an 8 week study period. Devices are preset to follow a scheduled activation pattern during the day.

SUMMARY:
To determine the extent to which the Apollo System is effective in reducing symptomatology associated with ADHD.

DETAILED DESCRIPTION:
The objective of this project is to understand the potential therapeutic benefits of the Apollo System for children with ADHD. Using vibrational therapy, the Apollo System has been previously demonstrated to promote greater balance of the autonomic nervous system. Given the importance of the autonomic nervous system for modulating levels of physiological arousal and in-turn governing aspects of attention and self-regulation; a therapeutic approach to promote better balance of this system may be particularly beneficial for populations such as children with ADHD. Accordingly, using a double-blind randomized placebo-controlled design this investigation will assess the extent to which the Apollo System is effective in reducing symptomatology associated with ADHD.

ELIGIBILITY:
Inclusion Criteria: All individuals that agreed to participate will be selected on a first come, first serve basis. No individual will be turned down due to sex, race, or ethnicity. The following inclusion criteria exist for all participants:

1. Participants must be 8 years of age or older and under the age of 18.
2. Participants must have diagnosed or suspected Attention Deficit Hyperactivity Disorder (ADHD).
3. Participants must have one of the following: 1) on the same treatment plan for over a year with minimal symptom relieve or alleviation, 2) tried two or more treatment approaches but is unable to meet treatment goals, 3) taking medication but still has symptoms, or 4) unwanted or uncontrollable side effects related to the medication.
4. Participants must have normal or corrected-to-normal vision in order to complete the cognitive task.

Exclusion Criteria: The following exclusion criteria exist for all participants:

1. Lack of consent.
2. Participants cannot have started a new treatment within the last 30 days.
3. Participants cannot have a history of hydrocephalus, Autism Spectrum Disorder, Schizophrenia, Conduct disorder, Oppositional Defiant Disorder, active substance abuse, or be on a beta blocker.
4. Participants cannot have previously used the Apollo System.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2022-03-18 (Actual); Primary Completion 2024-08-15 (Estimated); Study Completion 2024-08-15 (Estimated)

PRIMARY OUTCOMES:
Change in ADHD symptomatology as assessed using the ADHD-5 Rating Scale | Prior to and following the 8 week study protocol period.
  At pre and posttest, the parents/guardians of participants will complete the ADHD-5 Rating Scale. The behaviors included in the survey are derived from the diagnostic criteria for ADHD established in the Diagnostic and Statistical Manual of Mental Disorders, 5th edition. Scores are summated into inattentive and hyperactive-impulsive symptom domains and transformed into symptom percentile scores based upon normative data based on age and biological sex. Change in the overall ADHD percentile will be considered as the primary outcome. A more negative change would indicate a better outcome reflective of reduction in ADHD related symptomatology.
Effect Size for Change in Behavioral Index of Interference Control | Prior to and following the 8 week study protocol period.
  At pre and posttest, participants will complete a version of the Eriksen flanker task. Response accuracy will be quantified within each congruency as the proportion of correct responses relative to the number of trials administered. The effect size of the change from pre-to-posttest in overall response accuracy will be considered as the primary outcome.
  Effect sizes will be computed per Arm and do not reflect comparisons or combinations across Arms/Groups using the repeated measures variance correction for Cohen's d (Lakens, 2013).
Effect Size for Change in Behavioral Index of Response Inhibition | Prior to and following the 8 week study protocol period.
  At pre and posttest, participants will complete a version of the go/nogo task. Response accuracy will be quantified as the proportion of correct responses relative to the number of trials administered for target stimulus trails and nogo stimulus trials separately. The effect size of the change from pre-to-posttest for response accuracy to the nogo condition will be considered as the primary outcome.
  Effect sizes will be computed per Arm and do not reflect comparisons or combinations across Arms/Groups using the repeated measures variance correction for Cohen's d (Lakens, 2013).

CONTACTS AND LOCATIONS:
Overall Officials: Matthew B Pontifex, PhD., Principal Investigator — Michigan State University
Locations (1):
- Department of Kinesiology, East Lansing, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Data sharing will be by request and approval of the Michigan State University Human Research Protections Program with the provision of a data-safety and sharing agreement. No individually identifiable information will be shared.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available following primary publication of the results.
Access Criteria: By request and completion of an institutional data-safety and sharing agreement.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-19): https://cdn.clinicaltrials.gov/large-docs/06/NCT05308706/Prot_SAP_000.pdf